CLINICAL TRIAL: NCT04200716
Title: Evaluation of Vascular Responses to Moderate-intensity Continuous and High-intensity Interval Physical Exercise in Individuals With Prehypertension: a Randomized Trial
Brief Title: Arterial Function After Two Different Physical Exercise Intensities in Prehypertension
Acronym: PREHTEXVAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Luiz Aparecido Bortolotto, Director of Hypertension Unity Professor of Cardiology Department of Medical School São Paulo University, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 72503117.0.0000.0068; 165778/2017-2 (Other Grant/Funding Number: Conselho Nacional Desenvolvimento Científico e Tecnológico)
Record Dates: First submitted 2019-10-31; First posted 2019-12-16 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Prehypertension; Masked Hypertension
Keywords: Arterial function; Physical exercise; Arterial stiffness; Ambulatory Measurement of Blood Pressure
MeSH Terms: conditions — Prehypertension; Masked Hypertension; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate intensity continuous training - session (Active Comparator): The volunteers perform a 30-minute moderate-intensity exercise session on the exercise bike.
  Interventions: Behavioral: Moderate intensity continuous training - session; Behavioral: High intensity interval training - session
- High intensity interval training - session (Active Comparator): The volunteers perform a session of high intensity interval exercise on the exercise bike.
  Interventions: Behavioral: Moderate intensity continuous training - session; Behavioral: High intensity interval training - session

INTERVENTIONS:
Behavioral: Moderate intensity continuous training - session — Moderate exercise continuous exercise 30 minuts session
Behavioral: High intensity interval training - session — The high intensity interval exercise sessions are isocaloric to the moderate intensity continuous exercise, therefore, the necessary exercise time equivalent to 30 minutes of the moderate exercise continuous exercise session was calculated.

SUMMARY:
Individuals with prehypertension, diagnosed according to the 7th Brazilian Guidelines on Hypertension with the presence of systolic blood pressure (SBP) between 121 and 139 and / or diastolic (DBP) between 81 and 89 mmHg, are more likely to become hypertensive and to develop cardiovascular complications. Moreover, they already have alterations in the function of large arteries that may play a role in the development of the disease in the future. An option in the prevention / treatment of hypertension is the moderate intensity physical training, but high intensity interval training offers the possibility of greater exercise adherence, since it can be performed with less volume and less time spent, with the same benefits than moderate exercise, or even higher, being preferred by the population. Among these benefits, the investigators can mention the post-exercise hypotension (PEH) which occurs in normotensive, prehypertensive, and hypertensive individuals, due the decreased in sympathetic nerve activity and improved in vascular function. Also, selected participants with prehypertension can present a profile of masked hypertension, identified only by 24 hours ambulatory BP monitoring (ABPM). Given the possible differences between vascular responses to exercise intensities, the investigators intend to compare, in prehypertensive patients, the vascular responses of large arteries by noninvasive methods and PEH to a session of high intensity exercise and a session of moderate intensity continuous exercise. In addition, to study some of the possible physiological variables involved in this response by measuring heart rate variability. It is expected to find differences in vascular responses according to the presence of masked hypertension. Twenty two prehypertensive individuals aged between 30 and 60 years of both sexes will be studied. Subjects will perform cardiopulmonary testing and baseline vascular measurements (central pressure and pulse wave velocity measurements by three different methods), as well as 24 -hour ABPM. The vascular measurements will be repeated immediately after, and 24 hours after each session. Each participant will perform the session of one type of exercise in one day, and after three days will perform the other, with random distribution to the sequence of exercise type. Participants will perform 24-hour ABPM prior to exercise and for 24 hours after each exercise session. Data will be compared by appropriate statistical analysis.

DETAILED DESCRIPTION:
The measurement of central pressure and pulse wave velocity are achieved by three follow devices: Complior® , Sphygmocor® and Arteriograph®. The heart rate variability is achieved by Polar® device.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥30 and ≤60 years old
* Prehypertension, according to the 7 th Brazilian Arterial Hypertension Guideline values
* Both sexes
* Those who agree to sign the free and informed consent form

Exclusion Criteria:

* Engaged in other studies or programs of physical activity or training
* In drug treatment (for hypertension or other metabolic disease)
* Smokers
* Unable to perform exercise on exercise bike
* Presence of cardiovascular or metabolic disease (eg diabetes, hypercholesterolemia)
* Pregnant

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2018-07-03 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Changes in arterial stiffness by piezoelectric method (Complior) | Baseline, immediately after exercise and 24 hours after exercise
  Changes in arterial function behavior in response to two different physical exercise intensities.
Methods of measuring arterial stiffness: piezoelectric, tonometric and oscillometric | Baseline.
  Comparison of methods of evaluation of early markers of cardiovascular disease.

SECONDARY OUTCOMES:
Changes in heart rate variability | Baseline, immediately after exercise and 24 hours after exercise
  Changes in heart rate variability
Ambulatory systolic blood pressure measurement | During 24 hours after each exercise session
  Ambulatory measurement of 24-hours ambulatory systolic blood pressure
Ambulatory diastolic blood pressure measurement | During 24 hours after each exercise session
  Ambulatory measurement of 24-hours ambulatory diastolic blood pressure
Changes in arterial stiffness by three methods: piezoelectric, tonometric and oscillometric | Baseline, immediately after exercise and 24 hours after exercise.
  Changes in arterial function behavior in response to two different physical exercise intensities by three methods.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Bortolotto, Principal Investigator — Heart Institute (InCor), Hospital das Clinicas do HCFMUSP
Locations (1):
- Heart Institute (InCor), Hospital das Clinicas do HCFMUSP, São Paulo, Brazil

REFERENCES:
- [Derived] Rodrigues S, Verardino RGS, Costa-Hong V, Jordao CP, Jose Andrade da Costa M, Bortolotto L. Evaluation of vascular responses to moderate-intensity continuous and high-intensity interval physical exercise in subjects with elevated blood pressure: a randomised, cross-over clinical trial. Open Heart. 2025 Apr 2;12(1):e003121. doi: 10.1136/openhrt-2024-003121. PMID 40175098